CLINICAL TRIAL: NCT01315171
Title: The Effect of a Long-term Medium Chain Supplemented Diet on Cognitive Function and Brain Activation During Hypoglycemia in Type 1 Diabetes.
Brief Title: Effect of a Medium Chain Triglyceride Supplemented Diet on Cognitive Function and Brain Activation in Type 1 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1009007394
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Hypo-unawareness; Type 1 Diabetes Mellitus
Keywords: medium chain triglycerides; hypoglycemia; cognitive function; functional MRI
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medium chain supplemented diet (Experimental): Subjects will have a diet during which all meals are supplemented with 4 tablespoons of medium chain triglyceride oil.
  Interventions: Dietary Supplement: Medium chain triglycerides
- Standard group (No Intervention): Subjects will continue with a standard western diabetes diet.

INTERVENTIONS:
Dietary Supplement: Medium chain triglycerides — 4 tablespoons/day for 2 weeks
  Arms: Medium chain supplemented diet

SUMMARY:
Insulin treatment often causes the blood glucose levels to fall too low (hypoglycemia). Hypoglycemia can be associated with confusion and disorientation as well as other symptoms such as palpitations, sweating and tremors. Medium chain triglycerides (MCT) can be used as a fuel in the brain during low blood sugar levels and therefore may prevent or reduce some of the confusion and disorientation seen during hypoglycemia. We would like to determine if a diet supplemented with medium chain triglycerides can improve cognitive function during hypoglycemia, diabetes control and also look at brain activity.

DETAILED DESCRIPTION:
30 subjects with well controlled type 1 diabetes will be recruited for the study. If you agree to participate you will be scheduled for, dietitian visits, and a study visit which will include insulin and glucose infusions, an MRI scan and brain function tests. All visits will be on the Hospital Research Unit (HRU) on the 10th floor of Yale New Haven Hospital. You will be randomized to either the MCT-supplemented diet or the standardized western diabetic diet. If you are on the MCT diet, the MCT oil will be given to you and you will be shown how to incorporate it into your diet. The MCT supplemented diet is for two weeks (with a two gradual transition onto the diet) and the standardized western diet is for two weeks (with a 1 week transition onto the diet). At the end of the study you will be admitted to the Hospital Research Unit for the insulin 'clamp' and MRI scan. A 'clamp' is a procedure which involves insulin and glucose infusions. During a 'clamp' study, the insulin infusion is held constant, while the glucose infusion is adjusted every 5 minutes as needed to maintain the desired blood glucose levels. Compensation for the study is $750.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* HbA1c <8%
* BMI 18-30
* hypo unawareness

Exclusion Criteria:

* pregnancy
* significant diabetes complications
* liver disease, cirrhosis
* cardiac disease
* neurological disorder
* kidney disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2015-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cognitive function tests | 100 minutes
  Cognitive function will be assessed during hypoglycemia. 3 tests will be carried looking at working memory with number and word recollection.

SECONDARY OUTCOMES:
Brain activity | 100 minutes
  The fMRI will be used to assess brain activity during hypoglycemia in the presence of medium chain triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States